CLINICAL TRIAL: NCT03527043
Title: Assessing the Impact of Escitalopram on Sperm DNA Fragmentation: A Randomized Placebo Controlled
Brief Title: Impact of Escitalopram on Sperm DNA Fragmentation
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: funding stopped
Sponsor: Weill Medical College of Cornell University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1608017504
Record Dates: First submitted 2018-01-19; First posted 2018-05-16 (Actual); Results first posted 2025-03-25 (Actual); Last update posted 2025-08-06 (Actual); Status verified 2025-07

CONDITIONS: Sperm DNA Fragmentation; Infertility, Male
MeSH Terms: conditions — Infertility, Male | interventions — Escitalopram

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Escitalopram (Experimental): 10mg by mouth daily for 6 weeks
  Interventions: Drug: Escitalopram
- Placebo (Placebo Comparator): Matched placebo control by mouth for 6 weeks.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Escitalopram — 10mg by mouth daily for 6 weeks
  Arms: Escitalopram
Other: Placebo — matched placebo control by mouth for 6 weeks
  Arms: Placebo

SUMMARY:
Double-blind placebo-controlled randomized trial of daily escitalopram for 6 weeks in healthy men with normal semen analyses and no psychiatric history of depression, bipolar, mania or suicidal ideation. Hormone profiles, semen analysis, sperm DNA fragmentation, and sexual function will be measured at baseline, after 6 weeks of therapy, and 4 weeks after discontinuation of therapy (10 weeks into study).

DETAILED DESCRIPTION:
SSRI medications, specifically escitalopram is a very commonly prescribed medication among men of reproductive age. Significant evidence exists that they may be harmful for paternal fertility potential in both animal and human studies. However, high quality data is lacking, particularly among commonly used SSRI's such as escitalopram. As such, it is important to properly evaluate the potential effect of escitalopram in a randomized placebo controlled fashion. Results will be important in guiding urologists, psychiatrists and family practitioners regarding discussion surrounding SSRI use in their patients interested in fertility.

ELIGIBILITY:
Inclusion Criteria:

* Normal semen analyses, or semen analyses with at least 5 million sperm
* Normal TUNEL value (<7%)
* Willing to engage in at least weekly sexual activity, with a partner or alone for the duration of the 10-week study

Exclusion Criteria:

* Azoospermia or severe oligospermia (<5million sperm per semen analysis)
* Presently attempting to conceive pregnancy
* Sexual dysfunction preventing ability to provide semen analysis throughout study or engage in weekly sexual activity
* Current psychiatric disorder including: bipolar, mania, depression, generalized anxiety, social phobia, panic attacks, obsessive compulsive disorder, and schizophrenia.
* Family history of bipolar disorder, or suicide (including 2nd degree relatives)
* Present use of psychotropic agents (prescription or herbal) or anticonvulsants
* Use of sleeping pills
* Alcohol consumption greater that 2oz/day
* Use of illicit drugs
* Inability to read, follow instructions or complete questionnaires in English.
* Use of hormonal medications in past 3 months (androgens, androgen blockade, anabolic steroids, estrogens, herbal)
* Use of medications to enhance sexual function
* History of chemotherapy or pelvic radiation
* Use of Monoamine Oxidase inhibitors (MAOi's) or tricyclic antidepressants (TCAs) within 14 days
* Liver disease

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 75 (Actual)
Dates: Start 2017-10-01 (Actual); Primary Completion 2023-04-04 (Actual); Study Completion 2024-05-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan Gal, MD, Principal Investigator — Weill Medical College of Cornell University; Peter Schlegel, MD, Principal Investigator — Weill Medical College of Cornell University
Locations (1):
- Weill Cornell Medicine, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Escitalopram | Placebo
Started | 37 | 38
Completed | 36 | 38
Not Completed | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Escitalopram | Placebo | Total
Number analyzed (Participants) | 37 | 38 | 75
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 37 | 38 | 75
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 37 | 38 | 75
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 36 | 34 | 70
  Unknown or Not Reported | 1 | 4 | 5
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 5 | 1 | 6
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 17 | 16 | 33
  White | 11 | 12 | 23
  More than one race | 3 | 4 | 7
  Unknown or Not Reported | 1 | 4 | 5

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Patients Who Have Abnormal (>7%) TUNEL DNA Fragmentation Levels After 6 Weeks of Treatment
Description: TUNEL assay for sperm DNA fragmentation,Percentage of patients who have abnormal (>7%) TUNEL DNA fragmentation levels after 6 weeks of treatment
Time Frame: 6 weeks
Measure: Number; unit: Percentage
Arm/Group | Escitalopram | Placebo
Number analyzed (Participants) | 37 | 38
Percentage | 27 | 21.05

2. Secondary Outcome: Percentage of Patients Who Have Abnormal DNA Fragmentation Levels at 10 Weeks (4 Weeks Following Cessation of Treatment)
Description: Tunnel assay of the DNA fragmentation, Percentage of patients who have abnormal DNA fragmentation levels at 10 weeks (4 weeks following cessation of treatment)
Time Frame: 10 weeks
Measure: Number; unit: participants
Arm/Group | Escitalopram | Placebo
Number analyzed (Participants) | 37 | 38
participants | 24 | 18

3. Secondary Outcome: Absolute Change in DNA Fragmentation Percentage
Description: Absolute change in DNA fragmentation percentage across treatment groups from baseline
Time Frame: 0 (baseline), 6, 10 weeks
Measure: Mean (Standard Deviation); unit: Percentage
Arm/Group | Escitalopram | Placebo
Number analyzed (Participants) | 37 | 38
Percentage
  Baseline | 8.28 (5.61) | 7.2 (5.66)
  6 Weeks | 9.22 (7.23) | 8.3 (7.29)
  10 Weeks | 7.93 (7.05) | 7.39 (4.66)

4. Other Pre Specified Outcome: Serum Testosterone Measurement
Description: Change in serum testosterone (ng/dL)
Time Frame: 0 (baseline), 6, 10 weeks
Reporting Status: Not Posted

5. Other Pre Specified Outcome: Change in Serum Luteinizing Hormone (LH) (mIU/mL)
Description: Serum Luteinizing hormone measurement, Change in serum luteinizing hormone (LH) (mIU/mL)
Time Frame: 0 (baseline), 6, 10 weeks
Reporting Status: Not Posted

6. Other Pre Specified Outcome: Change in Serum Follicle-stimulating Hormone (FSH) (mIU/mL)
Description: Serum follicle-stimulating hormone measurement,Change in serum follicle-stimulating hormone (FSH) (mIU/mL)
Time Frame: 0 (baseline), 6, 10 weeks
Reporting Status: Not Posted

7. Other Pre Specified Outcome: Change in Serum Prolactin (ng/mL)
Description: serum prolactin measurement,Change in serum prolactin (ng/mL)
Time Frame: 0 (baseline), 6, 10 weeks
Reporting Status: Not Posted

8. Other Pre Specified Outcome: Change in International Index of Erectile Function Survey
Description: International Index of Erectile Function (IIEF) Survey. Severe Erectile Dysfunction (5-7), moderate (8-11), mild to moderate (12-16), mild (17-21), and no Erectile Dysfunction (22-25)
Time Frame: 0 (Baseline), 6, 10 weeks
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 10 weeks
Arm/Group | Escitalopram | Placebo
All-Cause Mortality (participants affected / at risk) | 0/37 | 0/38
Serious Adverse Events (participants affected / at risk) | 0/37 | 0/38
Other Adverse Events (participants affected / at risk) | 0/37 | 0/38

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-05-09): https://cdn.clinicaltrials.gov/large-docs/43/NCT03527043/Prot_SAP_000.pdf